CLINICAL TRIAL: NCT02313116
Title: Computed Optical Margin Assessment for Breast Cancer Surgery, Phase I (Part B)
Status: Suspended | Type: Observational
Sponsor: Diagnostic Photonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DxP 2012-02 (Part B)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Lumpectomy; Breast cancer; Optical coherence tomography; Tumor margin; Imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Interferometric Synthetic Aperture Microscopy — Optical coherence tomography with interferometric synthetic aperture microscopy will be used to image ex vivo breast tissue specimens.
  Other Names: Optical Coherence Tomography

SUMMARY:
This intraoperative study is a prospective study analyzing specimens from fifty subjects. Patients scheduled to undergo breast-conserving surgery will be recruited in accordance with the inclusion and exclusion criteria. The study period per subject is the time it takes to assess the ex vivo breast tissue sample using the study device. Image review will be conducted during surgery and compared to the margin status findings in the post-operative pathology report.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age or older
2. Signed informed consent form
3. Women who have been histologically diagnosed with carcinoma of the breast prior to surgery
4. Patients planning breast preservation and undergoing lumpectomy (partial mastectomy) procedure

Exclusion Criteria:

1. Multicentric disease (histologically diagnosed cancer in two different quadrants of the breast)
2. Neoadjuvant systemic therapy
3. All T4 tumors
4. Previous radiation in the operated breast
5. Prior surgical procedure in the same quadrant
6. Implants in the operated breast
7. Pregnancy
8. Lactation
9. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer undergoing lumpectomy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-02 (Estimated); Study Completion 2020-03-18 (Estimated)

PRIMARY OUTCOMES:
Patients With All Positive/Close Margins Correctly Identified With the Device | 1 week after surgery
Number of Margins With False Positive Device Readings | 1 week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Jacobs, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States